CLINICAL TRIAL: NCT06490419
Title: Effect of Ultrasound Cavitation Versus Electrolipolysis on Obese Infertile Women With Polycystic Ovarian Syndrome: a Randomized Controlled Trial
Brief Title: Effect of Ultrasound Cavitation Versus Electrolipolysis on Obese Infertile Women With Polycystic Ovarian Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Ahmed Hassan, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004229
Record Dates: First submitted 2024-06-30; First posted 2024-07-08 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electrolipolysis group (Experimental): The participants will be treated by electrolipolysis, in addition to the low-caloric diet of 1200 kcal/day.
  Interventions: Device: Electrolipolysis
- ultrasound cavitation group (Experimental): The participants will be treated by ultrasound cavitation, in addition to the low-caloric diet of 1200 kcal/day.
  Interventions: Device: ultrasound cavitation

INTERVENTIONS:
Device: Electrolipolysis — Hypocaloric diet:
  All patients were prescribed balanced hypocaloric diet (1200 kcal/day) by the nutrition specialist, with physiological nutrient content: carbohydrates-50%, proteins-20%, fats-30% and fiber daily consumption of 30 - 40 g in dry form (grain and vegetables). Calorie distribution: breakfast-40%, lunch-40%, dinner-20%. Behavioral therapy to correct eating disorders: diary of food and lifestyle, motivational phone calls every week
  Electrolipolysis:
  the participants will receive electrolipolysis applied to abdomen, thigh and gluteal regions, 3 sessions/week, for 3 months, 60 minutes/session; 30 minutes on the abdomen and thigh and 30 minutes on gluteal region. the device will be set to cause a contraction for 4 seconds followed by a relaxation for 4 seconds with a pulse width of 400 microseconds and a frequency of 20 pulses per minute.
  Arms: electrolipolysis group
Device: ultrasound cavitation — Hypocaloric diet:
  All patients were prescribed balanced hypocaloric diet (1200 kcal/day) by the nutrition specialist, as in the electrolipolysis group.
  ultrasound cavitation (UC): The participants will be treated by UC on the abdomen for 30 minutes, two sessions per week for 3 months. From standing position, the abdominal area of each patient will be divided transversally into 3 parts; part I: from the xiphoid process to 3 cm above the umbilicus, part II: from 3cm above the umbilicus to 2 cm below the umbilicus and part III: from 2 cm below the umbilicus to the pubic bone. Vertically, each part will be divided into right and left segments in relation to the linea alba, forming a total of 6 abdominal segments.
  The program of cavitation; frequency (40 kHz) will be chosen, the time will be adjusted at 30 minutes. The cavitational head will be, then, moved very slowly on each abdominal segment in a small circular movement for 5 minutes.
  Arms: ultrasound cavitation group

SUMMARY:
This study aims to determine the difference between the effect of ultrasound cavitation and electrolipolysis on obese infertile women with polycystic ovarian syndrome.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is the most prevalent endocrinopathy among women during reproductive age . PCOS affects 5-10% of women in reproductive age. It has an effect on quality of life , fertility and pregnancy.

Obesity plays a significant role in reproductive disorders, particularly in women. It is associated with anovulation, menstrual disorders, infertility, difficulties in assisted reproduction, miscarriage, and adverse pregnancy outcomes.

The treatment of obesity and infertility causes some harm to women, due to the danger of some operations and medications other than the high cost of these operations, so it is necessary to use a therapeutic alternative that is non invasive, with lower risk and lower cost.

Both ultrasound cavitation (UC) and electrolipolysis are non invasive modalities with many positive effects on obesity and PCOS outcomes. The effect of both the UC and electrolipolysis has been separately investigated in previous studies. Though, no studies were found to compare the effect of both modalities in the management of infertile women with PCOS. Therefore, this study will be conducted to explore the effect of UC versus electrolipolysis on infertile women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Infertile married PCOS women, diagnosed by Rotterdam criteria .
* Their ages will be ranged between 25-35 year old.
* Their BMI will be ranged from 30-40 kg/ m2.
* Their waist/hip ratio equal to or more than 0.85

Exclusion Criteria:

* Thyroid dysfunction (hypothyroidism).
* Chronic and/or systemic illnesses (e.g. diabetes mellitus, liver, renal respiratory failure and cardiovascular disorders).
* Malignant tumors.
* Tubal adhesions as well as uterine abnormalities.
* Skin diseases in the abdominal and gluteal regions.
* Conditions that may prevent the use of electrical stimulation.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Weight, height and BMI measurements | within 3 months
  Weight/ height scale will be used to measure the weight and height of all females in both groups to calculate their BMI before and after treatment according to the following equation BMI = weight/height2 (kg/ m2)
Waist hip Ratio | within 3 months
  To accurately measure central obesity, waist/hip ratio will be measured by tape measurement. Waist circumference will be measured at the narrowest portion of the torso approximately midway between the lower costal margin and the iliac crest. The hip circumference will be measured over the widest portion of the gluteal and greater trochanteric region then the ratio between them will be calculated. Reference of female measurements for central obesity will be a waist circumference of >88 cm and a waist-hip ratio >0.85.
LH/ FSH Ratio | within 3 months
  ELISA kites will be used for assessing serum luteinizing hormone (LH) and follicular stimulating hormone (FSH) to calculate LH/ FSH ratio. Blood samples will be drawn from antecubital vein of each patient before and after treatment. It will be centrifuged within 2 hours after withdrawal. Serum will be stared at -20°C and assayed for LH/ FSH Ratio. They will be measured in the third day of the menstrual cycle but will be measured in the luteal phase
Ovulation rate | within 3 months
  Abdominal ultrasongraphy will be used to assess ovarian volume before and after treatment for measuring ovulation rate. A minimum of 12 follicles with a diameter of 2 to 9 mm in each ovary, as well as a rising ovarian volume with a minimum size of 10 mm, are the criteria required for an ultrasound diagnosis of defective ovulation

CONTACTS AND LOCATIONS:
Overall Officials: Afaf Botla, PHD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol